CLINICAL TRIAL: NCT02914431
Title: A Randomized Controlled Trial of the Accuracy of Maxillary Repositioning Using Personalized Titanium Plates vs CAD/CAM Surgical Splints in Orthognathic Surgery
Brief Title: Personalized Titanium Plates vs CAD/CAM Surgical Splints in Maxillary Repositioning of Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, wang xu dong, Director of Department of Oral and Craniomaxillofacial Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20152225
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion; Abnormalities, Jaw
Keywords: Personalized Titanium Plate; Orthognathic Surgery; Maxilla Repositioning; Accuracy; Computer-aided Design and Manufacturing; Patient Specified Implants (PSI)
MeSH Terms: conditions — Malocclusion; Jaw Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Printing Personalized Titanium Plate (Experimental): After the LeFort I osteotomy, the intraoperative repositioning and fixation of the maxilla is accomplished using 3D printing personalized titanium plates.
  Interventions: Device: 3D Printing Personalized Titanium Plate
- CAD/CAM Surgical Splint (No Intervention): After the LeFort I osteotomy, the intraoperative repositioning of the maxilla is accomplished using CAD/CAM surgical splints and the fixation of the maxilla is accomplished using commercialization titanium plates.

INTERVENTIONS:
Device: 3D Printing Personalized Titanium Plate — The cutting guides were placed onto the planned position. The cutting guides also worked as the drilling guide. Several screw holes were drilled using the predetermined screw holes on the guides. The osteotomy / ostectomy then start. Next, the 3D printing personalized maxillary fixation plates were adapted to reposition the Le Fort I segment to the planned position. The screw holes on the bones prepared by the cutting guides were used as the bony reference. The personalized plate was first firmly installed on the maxilla above the osteotomy line by aligning the corresponding screw holes on the plate to the bone. Afterwards, the position of the osteotomized Le Fort I segment was adjusted till all the remaining corresponding screw holes on bone and plate were aligned.
  Arms: 3D Printing Personalized Titanium Plate

SUMMARY:
The purpose of this study is to determine whether personalized titanium plates can achieve better accuracy than CAD/CAM surgical splint in maxilla repositioning in orthognathic surgery, and evaluate the feasibility of this technique in clinical application.

DETAILED DESCRIPTION:
The repositioning of maxillary segment is essential for esthetic and functional outcomes in orthognathic surgery. With the giant leap in three-dimensional (3D) computer-aided surgical simulation (CASS) technology development, surgeons are now able to simulate various surgical plans in a computer to achieve the best possible outcome. In order to transfer the virtual surgical plan to the patient at the time of the surgery, surgical splints manufactured by computer-aided design and manufacturing (CAD/CAM) technique has been traditionally used to intraoperative reposition the maxilla. Nonetheless, the position of maxilla is still dependent to mandibular autorotation. The instability of the mandibular condyle-fossa relationship is a potential problem that may directly affect the placement of the maxillary segment at the desired position. Personalized titanium plates manufactured using titanium 3D printing technique have been used for maxilla repositioning and fixation to improve the operative accuracy in orthognathic surgery. Despite this, the evidence for advantage of this personalized titanium plates technique is not very strong and based on only a few studies.

The purpose of this study is to determine whether personalized titanium plates can achieve better accuracy than CAD/CAM surgical splint in maxilla repositioning in orthognathic surgery. The accuracy of using both methods for maxilla repositioning was quantitatively evaluated using linear and angular measurement. Secondary outcomes include operative time, amount of intraoperative blood loss, preoperative preparation time and treatment cost will also be measured to evaluate the feasibility of clinical application of personalized titanium plates technique in orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with skeletal dentofacial deformity and scheduled to undergo orthognathic surgery including maxillary surgery
* patients who were scheduled to undergo a computed tomography (CT) scan as a part of their diagnosis and treatment
* patients who agreed to participate in this study

Exclusion Criteria:

* Patients who had the previous orthognathic surgery
* Patients who had the previous maxillary or mandibular trauma
* Patients who had the maxillofacial tumor
* Patients who required the segmental maxillary surgery
* Oral soft tissues defect
* Within the infection period
* Craniofacial syndromes
* Bone metabolism disturbance
* Allergic to the titanium implant
* Unable to give informed consent
* Psychiatric disorders including dementia that may interfere with the study protocol
* Pregnancy
* Included in other studies
* Severe craniomandibular disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Difference of the maxillary position | 3 days after the operation
  Three landmark points (Upper dental midline between the 2 maxillary central incisal embrasure and both side mesiobuccal cusp of the upper 1st molar) were adopted on the maxilla, and the coordinates of these three landmarks were used to calculate the centroid of the maxilla. Positional differences of the centroid of the maxilla between the virtual plan and the actual result were measured.

SECONDARY OUTCOMES:
Intraoperative blood loss | Operative day
  Intraoperative blood loss
Operative time | Operative day
  Time cost of the operation
Translational differences of the maxilla | 3 days after the operation
  The translation differences of the centroid of the maxilla between the virtual plan and the actual result were calculated in X, Y and Z axis.
Orientational differences of the maxilla | 3 days after the operation
  The coordinates of all three landmarks of the maxilla was used to calculate the differences of orientation between the plan and postoperative results, which were calculated in pitch (the rotation around the X axis), roll (the rotation around the Y axis), and yaw (the rotation around the Z axis).

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Wang, MD, PhD, Study Director — Department of Oral and Craniomaxillofacial Surgery
Locations (1):
- Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No